CLINICAL TRIAL: NCT07339813
Title: Understanding Motor Function in Stroke Patients and Their Functional Brain Reorganization Using Ultra High-field MRI (MOTF-STROKE)
Brief Title: Understanding Motor Function in Stroke Patients and Their Functional Brain Reorganization Using Ultra High-field MRI
Acronym: MOTIF-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Principal Investigator, Myriam Edjlali-Goujon, Prof., Commissariat A L'energie Atomique
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEA 100 077
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: motor disability; functionnal MRI; High-field MRI; disconnection atlas; diffusion-weighted MRI; machine learning algorithms
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: RIPH 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic-Phase Ischemic Stroke Patients and Healthy Volunteer Optimization (Other): Participants undergo task-based and resting-state fMRI sessions. Imaging and clinical data are collected and analyzed using artificial intelligence models.
  Interventions: Other: Functional MRI (fMRI) Acquisition

INTERVENTIONS:
Other: Functional MRI (fMRI) Acquisition — Participants undergo task-based and resting-state fMRI sessions, including motor imagery and motor execution tasks. Brain activity and clinical data are collected for analysis.

SUMMARY:
The MOTIF-STROKE study is embedded within the BrainSync project, aiming to develop innovative strategies for motor rehabilitation of the upper limb. The primary goal is to construct a high-resolution anatomo-functional disconnection atlas in a cohort of 100 stroke patients, using cutting-edge 3T and 7T MRI. Data acquisition, commencing in Fall 2025, will combine morphological (T1-weighted), functional and diffusion-weighted MRI scans to perform morphometry, functional and structural connectivity analyses with biomarkers of motor deficits. This atlas seeks to correlate connectivity with motor tasks, using dedicated task-related fMRI paradigms and digital consultation tools. The project utilizes machine learning algorithms and functional hyper-alignment to analyze fMRI data, focusing on input features and their impact on prediction accuracy. The ultimate objective is to optimize implantation of WIMAGINE neuroprostheses for the subsequent BCI4STROKE clinical trial. Expected results include identifying clinical subgroups responsive to motor intention decoding, characterizing phenotypes of functional reorganization, and making the 3D brain atlas accessible to the neuroscience community.

ELIGIBILITY:
Inclusion Criteria:

Patients

* 1-MRI-confirmed diagnosis of a first ischemic stroke occurring more than 6 months prior to inclusion.
* 2-Persistent upper-limb motor deficit resulting from the stroke.
* 3-Absence of significant cognitive impairment: MMSE score ≥ 27 assessed as part of clinical care.
* 4-Age between 18 and 70 years.
* 5-Validation by the inclusion validation committee.
* 6-Signed informed consent after clear and fair information about the study.

Healthy volunteers:

* 1-Age between 18 and 70 years.
* 2-No history of neurological or psychiatric disease.
* 3-Signed informed consent after clear and fair information about the study.

Exclusion Criteria:

Patients:

* 1-Recurrent stroke.
* 2-Severe aphasia or severe speech disorders preventing adequate interaction for the protocol.
* 3-Severe auditory or visual impairment.
* 4-Disorders of comprehension, attention, or neglect affecting understanding of study motor tasks.
* 5-Associated conditions with an estimated life expectancy of less than 2 years.
* 6-History of brain surgery, craniectomy, or cranioplasty.
* 7-Other causes of motor disability.
* 8-Alcohol consumption the day before or on the day of the examination, or use of illicit psychotropic substances within 48 hours prior to MRI.
* 9-Absolute contraindications to MRI, including pregnancy; intracorporeal metallic foreign bodies; pacemakers; non-MRI-compatible neurostimulators; cochlear implants; implanted medical devices (electronic or non-electronic) implanted for less than 6 weeks; metallic heart valves; stents, coils, carotid or neurosurgical clips; implantable ports; infusion pumps; non-removable piercings; tattoos or permanent makeup larger than 5 cm on the head, neck, trunk, or upper limbs; transdermal devices with metallic components; intrauterine devices (except Mirena); dental appliances larger than 4 cm; or health conditions incompatible with MRI comfort and safety (e.g., acute respiratory or cardiac failure, inability to remain supine, bedridden state, claustrophobia).
* 10-Individuals not covered by a social security system.
* 11-Individuals under enhanced protection, including pregnant or breastfeeding women, persons deprived of liberty, legally protected adults, or patients in emergency situations.
* 12-Pregnant or breastfeeding women, or women of childbearing potential refusing a pregnancy test.

Healthy volunteer:

* 1-Absolute contraindications to MRI as listed above.
* 2-Individuals not covered by a social security system.
* 3-Individuals under enhanced protection, including pregnant or breastfeeding women, persons deprived of liberty, legally protected adults, or patients in emergency situations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Prediction accuracy of AI models for individual motor action intention | 1 day
  Validation of AI model predictions based on post-processing of functional MRI signals will be performed by comparing them with observed clinical performance during intentional motor tasks. These include assessment of movement intention of the hand and foot, intended movement direction, pathological side, and healthy side.

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Edjlali-Goujon, MD, PhD, Principal Investigator — Commissariat A L'energie Atomique
Locations (1):
- NeuroSpin, CEA, Gif-sur-Yvette, Île-de-France Region, France